CLINICAL TRIAL: NCT04951310
Title: COVID-19 Vaccinations With a Sweepstakes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Philadelphia Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 849044
Record Dates: First submitted 2021-06-16; First posted 2021-07-06 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Covid19
Keywords: COVID19 vaccination; Behavioral science interventions; Vaccination promotion
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No Intervention: Control participants (residents of Bucks County, Montgomery County, Delaware County, and Allegheny County, PA) are not eligible for the sweepstakes.
- Selected Zip Code Treatment (Experimental): Selected Zip Code Treatment participants will have a significantly greater chance to win a prize in the sweepstakes than all other Philadelphia residents. Half of all prizes in every drawing will go to Philadelphia residents in the selected zip code.
  Interventions: Behavioral: Philly Vax Sweepstakes
- All other Philadelphia Residents Treatment (Experimental): All other Philadelphia Residents Treatment participants will be eligible for the sweepstakes. Half of all prizes in every drawing will go to Philadelphia residents outside of the selected zip code.
  Interventions: Behavioral: Philly Vax Sweepstakes

INTERVENTIONS:
Behavioral: Philly Vax Sweepstakes — The "Philly Vax Sweepstakes" is a citywide sweepstakes designed to motivate Philadelphians to get vaccinated against COVID-19. A total of 36 vaccinated Philadelphians will win among three cash prize packages, distributed from the total cash pool. These 36 will be chosen over three drawings, with 12 residents chosen in each drawing.
  Arms: All other Philadelphia Residents Treatment; Selected Zip Code Treatment

SUMMARY:
To reach herd immunity for COVID-19, experts estimate that 70% of the population will need to be vaccinated. However, vaccination rates have begun to slow down in the United States. The investigators will partner with Philadelphia to launch a COVID-19 vaccination sweepstakes, in which residents will be eligible to win if they have received at least one dose of the COVID-19 vaccine prior to a given drawing. Drawings will be held every two weeks; multiple prizes of various sizes will be awarded in each drawing. Half of the prizes in each size category in each drawing will be awarded to residents of a zip code that is randomly selected from a pre-defined list of under-vaccinated zip codes (this zip code will be announced at the start of each 2-week drawing period), the other half will be awarded to residents outside of that selected zip code. The investigators will analyze vaccination rates in Philadelphia as compared with neighboring regions before, during, and after the specified time period, as well as analyze vaccination rates in the three selected zip codes compared to the other zip codes that could have been targeted (the residual set of under-vaccinated zip codes) to determine the effectiveness of the sweepstakes at encouraging vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* All 18+ residents of the City of Philadelphia will be eligible. Residents will be able to win the sweepstakes prizes if they can verify they received at least one dose of the COVID-19 vaccine before the date of the sweepstakes drawing in question.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3827656 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-08-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For our sweepstakes cash prizes, selected ZIP Codes with a high selection of cash prize winners (12 residents in each drawing) were 19126, 19133, and 19142 during Periods 1, 2, and 3, respectively.
Groups:
- Selected Zip Code Treatment: For our sweepstakes cash prizes, selected ZIP Codes with a high selection of cash prize winners (12 residents in each drawing) were 19126, 19133, and 19142 during Periods 1, 2, and 3, respectively.
- All Other Philadelphia Residents Treatment: Philadelphia has 46 residential zip codes. During each treatment period one of these zip codes was randomly chosen to be the selected zip code. The other 43 zip codes were therefore in the All other Philadelphia Residents Treatment.
Period: First Treatment Period (6/7/21-6/20/21)
Arm/Group | Control | Selected Zip Code Treatment | All Other Philadelphia Residents Treatment
Started | 2585846 | 52874 | 1188936
Completed | 2585846 | 52874 | 1188936
Not Completed | 0 | 0 | 0
Period: Second Treatment Period (6/21/21-7/5/21)
Arm/Group | Control | Selected Zip Code Treatment | All Other Philadelphia Residents Treatment
Started | 2585846 | 52874 | 1188936
Completed | 2585846 | 52874 | 1188936
Not Completed | 0 | 0 | 0
Period: Third Treatment Period (7/6/21-7/19/21)
Arm/Group | Control | Selected Zip Code Treatment | All Other Philadelphia Residents Treatment
Started | 2585846 | 52874 | 1188936
Completed | 2585846 | 52874 | 1188936
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Investigators did not collect demographic data as a part of this study. Instead, we used publicly available CDC data on the number of vaccinations per zip code.
Groups:
- Selected Zip Code Treatment: A total of 36 vaccinated Philadelphians won three cash prize packages, distributed from the total cash pool. These 36 were chosen over three drawings (i.e. treatment periods), with 12 residents chosen in each drawing. Selected Zip Code Treatment participants won half of these prizes and therefore had a significantly greater chance to win a prize in the sweepstakes than all other Philadelphia residents. A total of three zip codes were selected over the course of the Philly Vax Sweepstakes, one during each of the three treatment periods (19126 during period 1, 19133 during period 2, 19142 during period 3).
- Total: Total of all reporting groups
Arm/Group | Control | Selected Zip Code Treatment | All Other Philadelphia Residents Treatment | Total
Number analyzed (Participants) | 2585846 | 52874 | 1188936 | 3827656
Age, Customized [Count of Participants; unit: Participants] — Population: As the analysis population was all residents in target Philadelphia zip codes, demographic information including age was not available to investigators and was not collected as a part of this study.
Sex/Gender, Customized [Number; unit: participants] — Population: As the analysis population was all residents in target Philadelphia zip codes, demographic information including sex was not available to investigators and was not collected as a part of this study.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2585846 | 52874 | 1188936 | 3827656

OUTCOME MEASURES:

1. Primary Outcome: Weekly Vaccinations Per 100k Residents
Description: The primary outcome is the weekly vaccinations (per 100k residents) for residents receiving a first dose of a COVID-19 vaccination in each zip/county/city, relative to the control group. The vaccination data was measured by local health departments and the residency data was measured by the U.S. Census. The investigators included data from 5 weeks of pre-intervention, 6 weeks of intervention, and 4 weeks of post-intervention. Weekly Vaccinations per 100k Residents = 100,000 * Total residents receiving a first dose that week / Total residents in that zip/county/city code as measured by the Census or other official sources, at the most recent date available for all geographies of interest.
Time Frame: 15 Weeks
Measure: Number; unit: Weekly Vaccinations per 100k Residents
Arm/Group | Control | Selected Zip Code Treatment | All Other Philadelphia Residents Treatment
Number analyzed (Participants) | 2585846 | 52874 | 1188936
Weekly Vaccinations per 100k Residents | 0 | -4 | 383

ADVERSE EVENTS:
Time Frame: 6 weeks during the lottery period, from 6/7/21 until 7/19/21.
Arm/Group | Control | Selected Zip Code Treatment | All Other Philadelphia Residents Treatment
All-Cause Mortality (participants affected / at risk) | 0/2585846 | 0/52874 | 0/1188936
Serious Adverse Events (participants affected / at risk) | 0/2585846 | 0/52874 | 0/1188936
Other Adverse Events (participants affected / at risk) | 0/2585846 | 0/52874 | 0/1188936

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT04951310/Prot_SAP_000.pdf